CLINICAL TRIAL: NCT06837233
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase IIb/III Study to Assess the Efficacy and Safety of PG-011 Nasal Spray in Adults With Moderate to Severe Seasonal Allergic Rhinitis
Brief Title: A Study to Assess the Efficacy and Safety of PG-011 Nasal Spray in Adults With Moderate to Severe Seasonal Allergic Rhinitis
Acronym: Pumecitinib
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Prime Gene Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PG-011-SAR-301; CTR20250489 (Other: China's National Medical Products Administration (NMPA)，http://www.chinadrugtrials.org.cn/index.html)
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: SAR; PG-011; Seasonal Allergic Rhinitis; Pumecitinib
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PG-011 nasal spray 0.3% (twice daily) (Experimental): 2 sprays in each nostril, twice daily for 14-day treatment period.
  Interventions: Drug: Pumecitinib Nasal Spray 0.3%
- PG-011 nasal spray 0.6%(once daily) (Experimental): 2 sprays in each nostril, once daily for 14-day treatment period.
  Interventions: Drug: Pumecitinib Nasal Spray 0.6%; Drug: Placebo
- PG-011 nasal spray 0.6%(twice daily) (Experimental): 2 sprays in each nostril, twice daily for 14-day treatment period.
  Interventions: Drug: Pumecitinib nasal spray 0.6%(twice daily)
- Vehicle nasal spray(twice daily) (Placebo Comparator): 2 sprays in each nostril, twice daily for 14-day treatment period.
  Interventions: Drug: Placebo (twice daily)

INTERVENTIONS:
Drug: Pumecitinib Nasal Spray 0.3% — 2 sprays in each nostril, twice daily for 14-day treatment period.
  Arms: PG-011 nasal spray 0.3% (twice daily)
Drug: Pumecitinib Nasal Spray 0.6% — 2 sprays in each nostril, once daily for 14-day treatment period.
  Arms: PG-011 nasal spray 0.6%(once daily)
Drug: Placebo (twice daily) — 2 sprays in each nostril, twice daily for 14-day treatment period.
  Arms: Vehicle nasal spray(twice daily)
Drug: Pumecitinib nasal spray 0.6%(twice daily) — 2 sprays in each nostril, twice daily for 14-day treatment period.
  Arms: PG-011 nasal spray 0.6%(twice daily)
Drug: Placebo — 2 sprays in each nostril, once daily for 14-day treatment period.
  Arms: PG-011 nasal spray 0.6%(once daily)

SUMMARY:
The study is a multicenter, randomized, double-blind, placebo-controlled seamless and adaptive-designed phase IIb/III study encompassing a phase IIb and a phase III component. The phase IIb study, which is registered this time, is a dose-ranging component. The phase III study is a pivotal part of the overall research.

The goal of this phase IIb study is to evaluate the efficacy, safety, and pharmacokinetics of PG-011 nasal spray across various dosages and administration frequencies for treating adults with moderate to severe seasonal allergic rhinitis (SAR). Investigators will compare PG-011 nasal spray to a placebo (a look-alike substance that contains no drug) to see which dosage and frequency works to treat moderate to severe seasonal allergic rhinitis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled clinical study in adults participants aged from 18 to 65 years old (including threshold) with moderate to severe SAR. Approximately 160 participants will be randomized assigned to one of the 4 following groups in a 1:1:1:1 ratio.

PG-011 nasal spray 0.3% ( 0.6mg Pumecitinib) administered twice daily, PG-011 nasal spray 0.6% (1.2mg Pumecitinib) administered once daily, PG-011 nasal spray 0.6% (1.2mg Pumecitinib) administered twice daily, PG-011 placebo nasal spray 0% (0 mg Pumecitinib) administered once or twice daily.

Participants will receive blinded study treatment for 14 days followed by 21 days safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 65 (including threshold).
2. Reflective total nasal symptom score ( rTNSS) score≥ 6 and retrospective nasal obstruction ≥ 2 on the day of screening visit, D-4 and D1. Meanwhile, the baseline average rTNSS score(Calculated as the average of rTNSS score of D-3, D-2, D-1 morning, D-1 evening, and D1 morning) ≥ 6
3. History of SAR for at least 2 years. and positive results for any local allergen in the current season tested by either the skin prick test (SPT) (where the wheal diameter is at least 5 mm larger than that of the negative control) or the serum - specific IgE (sIgE) test (the sIgE test results obtained within ≤ 1 year before random enrollment are acceptable).
4. Willingness to avoid pregnancy or fathering children from the signing of the informed consent form until one month after the last administration of the investigational medicinal product.
5. Willing to sign the informed consent form and abide by the research protocol.

Exclusion Criteria:

1. Participants are diagnosed of active or latent tuberculosis infection.
2. Participants are diagnosed of moderate to severe asthma.
3. Participants who had active pulmonary diseases or infections (including but not limited to bronchitis, pneumonia), upper respiratory tract infections or sinus infections within 4 weeks before screening, and/or those who had respiratory infections during the lead-in period.
4. Participants received nasal or sinus surgery within 3 months before screening or had nasal trauma that had not fully healed.
5. Any nasal mucosal erosion, nasal septal ulcer, nasal septal perforation or other nasal diseases that, as judged by the investigator, may affect the deposition of drugs in the intranasal, such as acute or chronic sinusitis, drug-induced rhinitis, nasal polyps, etc.
6. Participants has ocular herpes simplex or other ocular infections (except seasonal allergic conjunctivitis).
7. Participants with facial or systemic fungal, bacterial, viral or parasitic infections, or oral infections that had not been cured and still required continuous treatment within 4 weeks before screening.
8. Participants have severe diseases such as central nervous system, respiratory system, liver, kidney, gastrointestinal tract, urinary system, endocrine system or blood system, which may affect the judgment of efficacy and safety .
9. Participants who were infected with human immunodeficiency virus (HIV) at the time of screening, those in the active stage of hepatitis C virus (HCV) infection (anti - HCV positive), those in the active stage of hepatitis B virus (HBV) infection (HBV - DNA > 2000 IU/mL or 10⁴ copies/mL), or those with positive Treponema pallidum antibody indicating an active stage of infection.
10. Any drug treatments before lead-in period, such as use of nasal or systemic decongestants and anticholinergic drugs within 3 days, use of antihistamines such as cetirizine, fexofenadine, and loratadine within 5 days, systemic use of glucocorticoids within 4 weeks, or local use of glucocorticoids, mast cell stabilizers, tricyclic antidepressants, and leukotriene receptor antagonists within 2 weeks, and use of anti - allergic Chinese herbal medicines within 2 weeks.
11. During the trial, participants who cannot stop using JAK inhibitors, tricyclic antidepressants, glucocorticoids, decongestants, antihistamines (except loratadine, which is a rescue drug required during the treatment), leukotriene receptor antagonists, mast cell stabilizers (including sodium cromoglycate, nedocromil sodium, tetrazolium chromone, nedocromil sodium, pemirolast potassium, and tranilast, etc.), anticholinergic drugs, anti - allergic Chinese herbal medicines, and those who cannot stop using nasal irrigation.
12. Participants who have undergone desensitization therapy or received immunotherapy within 6 months prior to screening.
13. Participants who are known or judged by the investigator to potentially have an allergic reaction to the active ingredients or excipients of the investigational drug.
14. Participants who have a history of intolerance to intranasal administration.
15. Participants who plan to travel outside the local area for 2 consecutive days or more during the trial.
16. Participants who have participated in other clinical studies of investigational drugs or medical devices within 3 months prior to screening.
17. Participants who have a history of drug abuse or alcoholism within 1 year prior to screening
18. Female participants who are breastfeeding or pregnant at the time of screening
19. Reproductive - age participants (male or female) who plan to become pregnant, breastfeed, or donate sperm/eggs during the study or within 1 month after the study ends
20. Any other condition that, in the opinion of the investigator or sponsor, makes the subject unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in average retrospective Total Nasal Symptom Score (rTNSS) over the 14-day treatment period | Baseline and Day 14
  The reflective Total Nasal Symptom Score (rTNSS) was assessed by 12-hour reflective scoring (AM, PM) of the severity of four nasal symptoms (rhinorrhea, sneezing, nasal congestion, nasal itching). Scores ranged from 0 (no signs/symptoms evident) to 3 (severe signs/symptoms that is hard to tolerate). The rTNSS was calculated as the sum of the subject-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate). Higher scores indicate more severe nasal symptoms, while lower scores indicate less severe nasal symptoms.

SECONDARY OUTCOMES:
Percent change from baseline in average retrospective Total Nasal Symptom Score (rTNSS) over the 14-day treatment period | Baseline and Day 14
  The reflective Total Nasal Symptom Score (rTNSS) was assessed by 12-hour reflective scoring (AM, PM) of the severity of four nasal symptoms (rhinorrhea, sneezing, nasal congestion, nasal itching). Scores ranged from 0 (no signs/symptoms evident) to 3 (severe signs/symptoms that is hard to tolerate). The rTNSS was calculated as the sum of the subject-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate). Higher scores indicate more severe nasal symptoms, while lower scores indicate less severe nasal symptoms.
  Percent change is calculated as (Change from baseline / Baseline result *100).
Change and percent change from baseline in average instantaneous Total Nasal Symptom Score (iTNSS) over the 14-day treatment period | Baseline and Day 14
  The instantaneous Total Nasal Symptom Score (iTNSS) was assessed by instantaneous symptom severity of four nasal symptoms (rhinorrhea, sneezing, nasal congestion, nasal itching). Scores ranged from 0 (no signs/symptoms evident) to 3 (severe signs/symptoms that is hard to tolerate).The iTNSS was calculated as the sum of the subject-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate). Higher scores indicate more severe nasal symptoms, while lower scores indicate less severe nasal symptoms.
  Percent change is calculated as (Change from baseline / Baseline result *100).
Change and percentage change from baseline in average retrospective Ocular Symptom Total Score (rTOSS) over the 14-day treatment period | Baseline and Day 14
  The reflective Ocular Symptom Total Score (rTOSS) was assessed by 12-hour reflective scoring (AM, PM) of the severity of three rocular symptoms (itching/burning, tearing/watering, and redness).Scores ranged from 0 (no signs/symptoms evident) to 3 (severe signs/symptoms that is hard to tolerate). . The Total Ocular Symptom Score (TOSS) ranged from 0 to 9. Higher scores indicate more severe ocular symptoms, while lower scores indicate less severe ocular symptoms.
  Percent change is calculated as (Change from baseline / Baseline result *100).
Change and percent change from baseline in average instantaneous ocular symptom score (iTOSS) over 14-day treatment period | Baseline and Day 14
  The instantaneous Total ocular Symptom Score is a scale used to measure ocular symptom severity based on how the participant was feeling just before taking each dose of study medication. Scores ranged from 0 to 9, and calculated as the sum of participant's scoring of three individual ocular symptoms (itching/burning, tearing/watering, and redness) on a 0 to 3 categorical severity scale (0=absent, 1=mild, 2=moderate, and 3=severe).
  Percent change is calculated as (Change from baseline / Baseline result *100).
Change from baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) score of general activities on day 15 | Baseline and Day 15
  Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) has 28 questions in 7 domains (activity limitation, sleep problems, nose symptoms, eye symptoms, non-nose/eye symptoms, practical problems and emotional function). Each question on a 7-point scale (0 = not impaired at all - 6 = severely impaired). The overall RQLQ score is the mean of all 28 responses.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Professor, Principal Investigator — Beijing Tongren Hospital
Locations (20):
- China (20):
  - Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - Luo Yang First People's Hospital, Luoyang, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Baotou Central Hospital, Baotou, Neimenggu
  - Chifeng Municipal Hospital, Chifeng, Neimenggu
  - Shandong Second Provincial People's Hospital, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Yantai YuHuangDing Hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Linfen Central Hospital, Linfen, Shanxi
  - Linfen People's Hospital, Linfen, Shanxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi

IPD SHARING:
Plan to Share IPD: No